CLINICAL TRIAL: NCT05125887
Title: Remote Assessment of Outpatient With SARS-CoV-2
Brief Title: Remote Assessment of Outpatient With Severe Acute Respiratory Syndrome (SARS-CoV-2)
Acronym: EVIDENCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI21_0033/Evidence
Record Dates: First submitted 2021-11-11; First posted 2021-11-18 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Patients diagnosed positive for COVID on an outpatient basis will respond to a questionnaire by mail, at 24 month of diagnosis. This questionnaire will make it possible in particular to collect intercurrent events (hospitalization, emergencies, etc.).

SUMMARY:
Outpatient management of patients with a milder form of COVID may be associated to an unfavorable initial or deferred course in relation to the pathology.. Outpatients represent the bulk of patients with COVID-19. To know their evolution, their secondary complications and identifying a profile of "at risk" patients is essential for the prevention and care of future non-hospitalized patients, in an epidemic context still active.

This study could make it possible to redefine the follow-up of outpatients. The study consists of a simple questionnaire and possibly a teleconsultation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a PCR (polymerase chain reaction assay ) positive for Sars-COV-2 between the start of the pandemic and May 11, 2020
* Outpatient care
* Inclusion 24 months from the date of diagnosis of Sars-COV-2 (± 6 months)

Exclusion Criteria:

* Patients in EHPAD (accommodation facilities for dependent elderly people), home, retirement home, center for disabled people
* Patients under protective measure, curators or guardianship
* Patients with a pathology or condition that does not allow them to express their wishes
* Patients hospitalized when performing PCR or within 10 days with Sars-COV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had a positive PCR (polymerase chain reaction assay ) meeting the eligibility criteria could be included
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-12 (Estimated); Study Completion 2023-06-12 (Estimated)

PRIMARY OUTCOMES:
Medical procedures | At month 24
  number of medical procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Médecine Interne A, Limoges, France

IPD SHARING:
Plan to Share IPD: No